CLINICAL TRIAL: NCT04058860
Title: Study of Microcirculation During Extracorporeal Circulation in Cardiac Surgery; Challenging Near-infrared Spectroscopy With Microvascular Density and Metabolic Parameters
Brief Title: Study of Microcirculation During Extracorporeal Circulation in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Kyriakos Anastasiadis, Professor of Cardiac Surgery, AHEPA University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AHEPA_CTS
Record Dates: First submitted 2019-08-12; First posted 2019-08-16 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Heart Diseases
Keywords: Microcirculation; Cardiac Surgery
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: Patients undergoing open heart surgery with minimal invasive extracorporeal circulation (MiECC) according to accepted indications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Patients (Other): Patients undergoing open heart surgery with minimal invasive extracorporeal circulation (MiECC) according to accepted indications
  Interventions: Device: NIRS monitoring; Device: Cox monitoring; Device: Sublingual microscopy

INTERVENTIONS:
Device: NIRS monitoring — Cerebral and somatic near-infrared spectroscopy (rScO2) measurements
Device: Cox monitoring — Cerebral autoregulation monitoring
Device: Sublingual microscopy — Sublingual mucosal microcirculation measurements during surgery using side dark field (SDF) imaging

SUMMARY:
The aim of the proposed study is to evaluate microcirculatory alterations in patients undergoing open heart surgery under extracorporeal circulation. Positive clinical results evidenced with goal-directed perfusion and cerebral oximetry monitoring could be attributed to preserved microcirculation at tissue level.

DETAILED DESCRIPTION:
The aim of the proposed study is to evaluate microcirculatory alterations in patients undergoing open heart surgery under extracorporeal circulation. Microcirculatory changes during cardiac surgery have been investigated mainly during coronary procedures using the conventional extracorporeal circulation. There is no single study in the literature investigating microcirculatory alterations using a perioperative strategy of "physiologic" perfusion. Positive clinical results evidenced with goal-directed perfusion and cerebral oximetry monitoring could be attributed to preserved microcirculation at tissue level.

All patients will follow the same anaesthetic and perfusion protocol. The protocol for the evaluation of microcirculation will be based on:

* Cerebral near-infrared spectroscopy (rScO2) measurements (INVOS, Covidien-Medtronic Inc.).
* NIRS-Based Cerebral Autoregulation Monitoring: Analog arterial blood pressure signals will be digitized and then processed with the digital NIRS signals using a personal computer and a special ICM software (University of Cambridge, Cambridge, UK). Monitoring cerebral autoregulation ensures adequate renal perfusion. Hence, brain can be used not just as a target but also as an index organ indicating adequacy of perfusion.
* Somatic near-infrared spectroscopy (rSsO2) measurements (INVOS, Covidien-Medtronic Inc.).
* Sublingual mucosal microcirculation measurements during surgery using side dark field (SDF) imaging (MicroScan, Microvision Medical, Amsterdam, The Netherlands).

All measurements will be performed at the following time points:

T0: after induction of anaesthesia T1: after initiation of cardiopulmonary bypass T2: 10 minutes after cross- clamping the aorta T3: 10 minutes before removing the aortic cross-clamp T4: after weaning from extracorporeal circulation

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 and < 85 years with coronary artery disease and/or aortic valve disease undergoing open heart surgery with accepted indications

Exclusion Criteria:

* patients undergoing emergency surgery
* patients in preoperative cardiogenic shock with evidence of tissue malperfusion
* patients > 85 years of age
* patients with severe peripheral vascular disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of microcirculation | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Correlation of NIRS values with tissue microvascular activity

SECONDARY OUTCOMES:
Global perfusion | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Global perfusion using cerebral NIRS during extracorporeal circulation
Cerebral autoregulation | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Calculation of cerebral oximetry index (COx)
Goal-directed perfusion | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Correlation of goal-directed perfusion with microvascular capillary density during extracorporeal circulation
Somatic perfusion | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Peripheral tissue oxygenation as measured with somatic NIRS

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, MD, PhD, Principal Investigator — Cardiothoracic Department, AHEPA University Hospital, Thessaloniki, Greece; Helena Argiriadou, MD, PhD, Principal Investigator — Cardiothoracic Department, AHEPA University Hospital, Thessaloniki, Greece
Locations (1):
- Cardiothoracic Department, AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anastasiadis K, Antonitsis P, Deliopoulos A, Argiriadou H. A multidisciplinary perioperative strategy for attaining "more physiologic" cardiac surgery. Perfusion. 2017 Sep;32(6):446-453. doi: 10.1177/0267659117700488. Epub 2017 Mar 10. PMID 28692337
- [Background] Anastasiadis K, Antonitsis P, Ranucci M, Murkin J. Minimally Invasive Extracorporeal Circulation (MiECC): Towards a More Physiologic Perfusion. J Cardiothorac Vasc Anesth. 2016 Apr;30(2):280-1. doi: 10.1053/j.jvca.2016.01.018. Epub 2016 Jan 13. No abstract available. PMID 27013118
- [Background] Murkin JM. Cerebral oximetry: monitoring the brain as the index organ. Anesthesiology. 2011 Jan;114(1):12-3. doi: 10.1097/ALN.0b013e3181fef5d2. No abstract available. PMID 21178667
- [Background] Murphy GS, Hessel EA 2nd, Groom RC. Optimal perfusion during cardiopulmonary bypass: an evidence-based approach. Anesth Analg. 2009 May;108(5):1394-417. doi: 10.1213/ane.0b013e3181875e2e. PMID 19372313
- [Background] Koning NJ, Vonk AB, Meesters MI, Oomens T, Verkaik M, Jansen EK, Baufreton C, Boer C. Microcirculatory perfusion is preserved during off-pump but not on-pump cardiac surgery. J Cardiothorac Vasc Anesth. 2014 Apr;28(2):336-41. doi: 10.1053/j.jvca.2013.05.026. Epub 2013 Oct 23. PMID 24161555
- [Background] Kara A, Akin S, Ince C. The response of the microcirculation to cardiac surgery. Curr Opin Anaesthesiol. 2016 Feb;29(1):85-93. doi: 10.1097/ACO.0000000000000280. PMID 26658179
- [Background] den Uil CA, Lagrand WK, Spronk PE, van Domburg RT, Hofland J, Luthen C, Brugts JJ, van der Ent M, Simoons ML. Impaired sublingual microvascular perfusion during surgery with cardiopulmonary bypass: a pilot study. J Thorac Cardiovasc Surg. 2008 Jul;136(1):129-34. doi: 10.1016/j.jtcvs.2007.10.046. Epub 2008 May 2. PMID 18603065